CLINICAL TRIAL: NCT00380991
Title: Dermatological Evaluation of Topic Compatibility (Primary and Accumulated Dermical Irritability and Dermical Sensitivity) of Dermacyd Delicata (New Fragrance)
Brief Title: Topic Compatibility Dermacyd Delicata - New Fragrance - Lactoserum - Hygiene
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LACTO_L_01840
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Hygiene
MeSH Terms: interventions — lactoserum

INTERVENTIONS:
Drug: lactoserum

SUMMARY:
The purpose of this study is to demonstrate the absence of potential irritation (primary dermic irritability and cumulated dermic irritability) and allergy (sensibilization) of the product Dermacyd Delicata (new fragrance of Dermacyd)

ELIGIBILITY:
Inclusion Criteria:

* Phototype Skin I,II, III and IV
* Integral skin test in the region;

Exclusion Criteria:

* Lactation or gestation
* Use of Antiinflammatory and/or immunosuppression drugs
* Personal history of atopy;
* History of sensibilization or irritation for topic products;
* Active cutaneous disease;
* Use of new drugs or cosmetics during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50
Dates: Start 2006-05

PRIMARY OUTCOMES:
score evaluation of the cutaneous reaction, preconized by International Contact Dermatitis Research Group (ICDRG)

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-aventis, São Paulo, Brazil